CLINICAL TRIAL: NCT03382613
Title: Quantify Use of Anticoagulation to Improve Management of AF
Brief Title: A Study to Quantify Use of Anticoagulation to Improve Management of Atrial Fibrillation
Acronym: QUANTUM AF
Status: Terminated | Type: Observational
Why Stopped: Operating Company decided to stop study due to strategic realignment and budgetary reasons
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108407; NOPRODAFL0001 (Other: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Quality Improvement (QI) Program: Hospitals assigned to the QI program arm will begin the 4-month Preparatory Phase which is designed to introduce the institutional baseline reporting tools and materials related to performance improvement, and gain insight into their gaps in treatment, followed by 15 month Implementation Phase, which will consist of education, process, and engagement activities that are targeted at the hospital and healthcare provider level and then the Measurement Period at which time hospitals will complete a final survey to document specific interventions that were successfully implemented and perform a final retrospective chart review on selected patients.
- Usual Care: Hospitals assigned to the Usual Care arm will not participate in the structured QI program but will continue with their standard hospital practice in treating patients with atrial fibrillation (AF) at risk for ischemic stroke. Hospitals will also complete a final survey and final retrospective chart reviews during the Measurement Period.

SUMMARY:
The purpose of this study is to evaluate the impact of a hospital quality improvement (QI) program on the use of guideline-recommended oral anticoagulants (OAC) in hospitalized patients with atrial fibrillation (AF) at risk for ischemic stroke. Specifically, the study will determine whether the intervention, compared to Usual Care, will result in a greater increase in the proportion of patients with AF at risk for ischemic stroke who are appropriately treated with OAC.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient hospitalization
* Primary or secondary discharge International Classification of Diseases (ICD)-9/10 diagnosis code for AF paroxysmal (I48.0), persistent (I48.1), chronic (I48.2), or unspecified (427.31, I48.91)
* Proxied Congestive Heart failure (CHA2DS2-VASC) score greater than or equal to (>=) 2 using ICD-9 diagnosis scoring algorithm developed previously. The scoring algorithm will be expanded to include ICD-10 codes
* Discharged to home, skilled nursing facility, inpatient rehabilitation, or nursing home

Exclusion Criteria:

* Presence of artificial mechanical heart valve by ICD-9/10 diagnosis or procedure code during comorbid identification period or current hospitalization
* Surgical procedure during hospitalization for open heart surgery, brain, or spine
* Intravenous heparin given on the day of discharge without warfarin/oral anticoagulant (OAC), antiplatelets, and/or aspirin
* History of left atrial appendage occlusion, including the Watchman device
* Any in-hospital (current hospitalization) bleeding identified by ICD-9/10 diagnosis codes

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with atrial fibrillation (AF) at risk for ischemic stroke will be included.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2017-12-29 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
Change in the Percentage of Patients Treated With OAC From Baseline to Final Collection Periods | Baseline up to 20 months
  The impact of a hospital quality improvement (QI) program on the use of guideline-recommended oral anticoagulants (OAC) in hospitalized patients with atrial fibrillation (AF) at risk for ischemic stroke will be evaluated by measuring change in the percentage of patients treated with OAC, from baseline to Final Collection Periods.

SECONDARY OUTCOMES:
Percentage of Patients Readmitted to the Same Hospital | Up to 20 months
  Percentage of patients readmitted to the same hospital for all-cause readmissions, stroke-related readmissions, cardiovascular (CV)-related readmissions, and bleeding- related readmissions will be evaluated.
Percentage of Patients who Received OAC by Hospital Characteristics Subgroups | End of study (Month 20)
  Use of OAC at the end of study by hospital characteristics subgroups (that is, patients care mix, infrastructure-bed size, staffing, academic status, location, urban/rural, provider) will be determined.
Effect of Tools Components of the QI Program on the use of OAC | End of study (Month 20)
  The effect of the educational process-based components of the QI program relative to the Usual Care arm on the use of OAC will be evaluated.
Effect of Degree of Engagement in the QI Program | End of study (Month 20)
  A performance dashboard will be implemented to aggregate and display performance data.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (62):
- United States (62):
  - Banner Thunderbird, Glendale, Arizona
  - Banner Desert Medical Center, Mesa, Arizona
  - Banner Baywood Medical Center, Mesa, Arizona
  - Banner Heart Hospital, Mesa, Arizona
  - Banner University Medical Center, Phoenix, Arizona
  - Banner Estrella, Phoenix, Arizona
  - Banner Boswell Medical Center, Sun City, Arizona
  - Banner Del Webb, Sun City West, Arizona
  - Banner University Medical Center - South (BUMC-S), Tucson, Arizona
  - Banner University Medical Center - Tucson (BUMC-T), Tucson, Arizona
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - AMITA Adventist Medical Center Bolingbrook, Bolingbrook, Illinois
  - AMITA Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - AMITA Adventist Medical Center Hinsdale, Hinsdale, Illinois
  - AMITA St. Alexius Medical Center, Hoffman Estates, Illinois
  - AMITA Adventist Medical Center La Grange, La Grange, Illinois
  - SSM Health Good Samaritan Hospital, Mount Vernon, Illinois
  - Ephraim McDowell Regional Medical Center, Danville, Kentucky
  - St. Agnes Hospital, Baltimore, Maryland
  - Borgess Medical Center, Kalamazoo, Michigan
  - Fremont Health Medical Center, Fremont, Nebraska
  - Penn Medicine - Princeton Health, Plainsboro, New Jersey
  - AtlantiCare, Pomona, New Jersey
  - Southside Hospital, Bay Shore, New York
  - Our Lady of Lourdes Hospital, Binghamton, New York
  - Long Island Jewish Forest Hills, Forest Hills, New York
  - Huntington Hospital, Huntington, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Med Ctr, New Hyde Park, New York
  - Lenox Hill Hospital, New York, New York
  - Long Island Jewish Valley Stream, Valley Stream, New York
  - Samaritan Medical Center, Watertown, New York
  - The Jewish Hospital - Mercy, Cincinnati, Ohio
  - Mercy Anderson Hospital, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Mercy St. Rita's Medical Center, Lima, Ohio
  - Mercy Lorain Regional Medical Center, Lorain, Ohio
  - Mercy St. Charles Hospital, Oregon, Ohio
  - University Hospitals Regional Hospitals, Richmond Heights, Ohio
  - Mercy Health St Vincent Medical Center, Toledo, Ohio
  - Mercy St. Anne Hospital, Toledo, Ohio
  - Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Saint Francis Hospital, Tulsa, Oklahoma
  - St. Luke's University Health Network, Allentown, Pennsylvania
  - St.Luke's University Health Network - St.Luke's Cardiology Associates, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center, Scranton, Pennsylvania
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania
  - AnMed Health, Anderson, South Carolina
  - Avera McKennan Hospital, Sioux Falls, South Dakota
  - Hendrick Medical Center, Abilene, Texas
  - Methodist Dallas Medical Center, Dallas, Texas
  - Methodist Charlton Medical Center, Dallas, Texas
  - Methodist Mansfield Medical Center, Mansfield, Texas
  - Methodist Richardson Medical Center, Richardson, Texas
  - Inova Alexandria Hospital, Alexandria, Virginia
  - Inova Health Care Services, Falls Church, Virginia
  - Riverside Regional Medical Center, Newport News, Virginia
  - St Marys Medical Center, Huntington, West Virginia
  - Monongalia County General Hospital Company, Morgantown, West Virginia